CLINICAL TRIAL: NCT02418897
Title: Does Abnormal Neuromuscular Junction Function Play a Role in the Pathogenesis of Motor Fatigue in Women With Multiple Sclerosis?
Brief Title: Role of Neuromuscular Junction Function in Motor Fatigue in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L15-098
Record Dates: First submitted 2015-04-07; First posted 2015-04-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; multiple sclerosis; neuromuscular junction; SFEMG
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This pilot study will evaluate for the presence of neuromuscular junction (NMJ) defect in women with motor fatigue in multiple sclerosis by Single Fiber Electromyography (SFEMG) using the concentric needle electrode.

DETAILED DESCRIPTION:
The investigators will recruit 20 women with multiple sclerosis (MS) and fatigue and 10 normal controls with no identified causes of fatigue (no history of thyroid disease, anemia, liver disease, kidney disease, myasthenia gravis, and no major fatigue inducing medications). We will include MS patients with fatigue severity scale of ≥5. Patients with sleep disorders or significant depression will be excluded based on history, Epworth Sleepiness scale, and Beck's Inventory of Depression Scale. The study will include two clinic visits and a one-study visit. After informed consent is obtained (English and Spanish forms will be available), the following will be done during the study visit 1:

* Neurological examination: Using handgrip dynamometer of the dominant hand.

  * Maximum voluntary isometric contraction force (MVIC) of the handgrip; two contractions of as long as 5 seconds each.
  * Single 30 seconds sustained maximal contraction of the handgrip to assess static fatigue.
  * Series of brief maximal contraction over 30 seconds, Contractions will be timed at one contraction per second.
* Expanded Disability Status Scale (EDSS
* Fatigue severity scale (FSS) and modified fatigue impact scale (MFIS)
* Epworth Sleepiness scale for screening for sleep disorders.
* Beck's Inventory of Depression Scale for screening for depression. Clinic visit 2: The clinic visit 2 will be conducted 5-30 days after the clinic visit 1
* Neurological examination: Using handgrip dynamometer of the dominant hand.

  * Maximum voluntary isometric contraction force (MVIC) of the handgrip; two contractions of as long as 5 seconds each.
  * Single 30 seconds sustained maximal contraction of the handgrip to assess static fatigue.
  * Series of brief maximal contraction over 30 seconds, Contractions will be timed at one per second.
* Fatigue severity scale (FSS) and modified fatigue impact scale (MFIS)

Study Visit 3:

Electromyography (EMG) and SFEMG (Single Fiber Electromyography) of the extensor digitorum communis muscle (forearm muscle) will be performed on all women with fatigue and healthy controls at the TTUHSC electrophysiology lab to evaluate for NMJ abnormalities. The mean consecutive difference (MCD) of 20 pairs of single muscle fiber potentials will be collected using SFEMG from each of the 20 women with multiple sclerosis and fatigue and will be compared to MCD of 200 pair potentials from our recruited 10 normal control subjects and also to the previously published normative data.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for MS Group (20 women)

1. Patients with relapsing remitting multiple sclerosis.
2. Age 18 to 65 years
3. Diagnosed with motor fatigue in multiple sclerosis > 6 weeks. Motor fatigue equates to muscle fatigue due to physical exertion and is alleviated with rest and associated with fatigability.
4. Has a fatigue severity scale score (FSS) of ≥5.
5. Ambulatory with Expanded Disability Status Scale score (EDSS) 1.5 -6.5.

Inclusion Criteria for Control Group (10 women)

1. Female with no history of multiple sclerosis and no complaint of fatigue
2. Age 18 to 65 years

Exclusion Criteria:

1. Patients with MS exacerbation or corticosteroid treatment within one month before the study.
2. Patients with history or current diagnosis of:

   * Untreated thyroid disease,
   * Untreated vitamin D deficiency,
   * pregnancy,
   * taking over the counter energy booster in the last 1 week,
   * taking medication that will improve the function of the neuromuscular junction (i.e. pyridostigmine, steroid, rituximab, mycophenolate mofetil, azathioprine),
   * myasthenia gravis,
   * symptoms or history of polyneuropathy involving the upper extremities,
   * myopathy,
   * symptoms or history suggestive of C7, C 8 radiculopathy,
   * motor neuron disease,
   * polio,
   * chronic inflammatory demyelinating polyneuropathy,
   * Guillain-Barre syndrome,
   * radial nerve palsy,
   * sleep disorders (Epworth Sleepiness scale> 10 ), or
   * significant depression ( Beck's Inventory of Depression Scale >17)
3. Taking major fatigue inducing medications. (e.g. Narcotics, and Sedatives)
4. Taking anticoagulation therapy. (e.g. warfarin and heparin)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with relapsing remitting multiple sclerosis (MS) with motor fatigue in MS > 6 weeks. Motor fatigue equates to muscle fatigue due to physical exertion and is alleviated with rest and associated with fatigability.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal Jitter. | 8 months
  Single fiber electromyography (SFEMG) is used to measure the variation between firing of adjacent muscle fibers and to detect prolonged abnormal jitter. The two criteria that the investigator will use to demonstrate abnormal neuromuscular Junction function are the 10% of pairs with abnormal jitter or abnormal mean jitter value of the 20 pairs . The 95% confidence limit of all individual measurements has been used as upper limit of what is considered normal. For extensor digitorum communis (EDC), the 95% confidence limit of jitter in individual pair mean consecutive difference (MCD) is 49 microseconds (MCD of individual pair is 30.6+/-9.2 micros) and the 95% confidence limit of jitter (mean MCD) per study is 38.1 microseconds (MCD per study is 30.7+/-3.7 micros).

SECONDARY OUTCOMES:
Score of fatigue (Fatigue severity scale (FSS) and modified fatigue impact scale (MFIS)) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Eldokla, MD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States